CLINICAL TRIAL: NCT05859919
Title: Conducting Clinical Trials of the Medicine "Rutan Tablets 0.1g" No. 10 in the Complex Therapy of the Viral Disease COVID-19
Brief Title: Conducting Clinical Trials of the Medicine "Rutan Tablets 0.1g" No. 10 in the Complex Therapy of COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Research Institute of Virology, Ministry of Health of the Republic of Uzbekistan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: C-И-45
Record Dates: First submitted 2023-05-15; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Patients With COVID-19
Keywords: COVID-19; SARS-CoV-2; Rutan
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The study will be a series of comparisons with two groups. The main group will receive the drug "Rutan 0.1".
  The control group will not be given the study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The main group receiving the drug "Rutan 0.1" and (Experimental): The main group will receive the drug "Rutan 0.1"
  Interventions: Drug: The drug "Rutan 0.1".
- The control group not receiving Rutan 0.1 (Other): The control group will not be given the study drug Rutan 0.1
  Interventions: Other: Basic treatment

INTERVENTIONS:
Drug: The drug "Rutan 0.1". — Active ingredient: (3,6-bis-O-galloyl-1,2,4-tri-O-galloyl-β-D-glucose). Active substance: "Rutan 0.1" 100mg. Excipients: potato starch, calcium stearate, lactulose.
  Other Names: Rutan
  Arms: The main group receiving the drug "Rutan 0.1" and
Other: Basic treatment — Basic treatment without the drug "Rutan 0.1".
  Arms: The control group not receiving Rutan 0.1

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of the registered drug Rutan 0.1 against SARS-CoV-2 in patients with COVID-19.

The main group (30 people) - patients with COVID-19 who are on inpatient treatment who were prescribed the drug Rutan 0.1, 1 tablet 2 times a day for 10 days.

The control group (27 people) - patients with COVID-19 who are hospitalized and received therapy according to the National Temporary Protocol for the management of patients with COVID-19.

DETAILED DESCRIPTION:
This study is a randomized, open-label, controlled trial to evaluate the safety and efficacy of a novel therapeutic agent, Rutan 0.1, in hospitalized adult patients diagnosed with COVID-19. The study will be a series of comparisons with two groups. The main group will receive the drug "Rutan 0.1". The control group will not be given the study drug. There will be continuous monitoring to stop the study due to futility, efficacy or safety. Because of the likelihood that the baseline standards for maintenance therapy may evolve/improve over time, safety and efficacy comparisons will adapt.

Randomization will be based on: Card system (the patient will be asked to choose one of two cards with the same drawings on the visible side, and after choosing, when turning over the cards, it will be determined which group the patient will be included) Patients of the main group (30 patients) will be prescribed Rutan 0.1 tablets, along with the therapy recommended at the time of the study. The course of treatment will be - on the first day, 1 tablet 3 times a day, in the following days - 1 tablet 2 times a day. The duration of the course of treatment is 10 days, with good tolerability of the drug.

The comparison group (27 patients) will receive the current recommended treatment at the time of the study without the use of investigational drug.

Screening failures are defined by participants who agreed to participate in a clinical trial but were not subsequently randomized to participate in the study. A minimum set of information about monitoring failures is required to ensure transparent reporting, compliance with the publication of the Consolidated Reporting Standards (CONSORT), and responses to regulatory requests. The minimum information includes demographics, monitoring failure details, eligibility criteria, and any serious adverse events (SAEs).

Discontinuation of participation/withdrawal of a participant means termination of participation in the study, and the remaining study procedures must be interrupted and replaced by another participant, as indicated in the study protocol. Any clinically significant changes in the patient's condition and/or laboratory values will be reported as an adverse event (AE) by the investigator. The researcher has the right to make changes or terminate the study.

ELIGIBILITY:
Inclusion Criteria:

1. Providing a signed and dated informed consent form.
2. Declared willingness to comply with all study procedures and availability during the study.
3. Man or woman over the age of 18.
4. Patients with PCR-confirmed COVID-19 with mild/moderate disease. U07.1.
5. Ability to take oral medications and willingness to adhere to the regimen.
6. For women of childbearing potential: use of highly effective contraceptives for at least 1 month before screening and agree to use such a method during study participation and for an additional 4 weeks after the end.
7. For men of reproductive potential: use condoms or other methods to ensure effective contraception with a partner.
8. Agree to adhere to the lifestyle principles throughout the study period.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Severe form of COVID-19 disease. U07.1.
3. Treatment with another investigational drug.
4. Individual intolerance to the drug.
5. The occurrence of any allergic reactions.
6. Weighting of the general state of health of the patient and the transition to a severe form of the disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Check the safety and effectiveness of the drug "Rutan 0.1" | The duration of the course of treatment is 10 days
  In the experimental group, on days 4-5 of hospitalization in the hospital after taking rutan 100 mg, the PCR indicators for covid 19 were negative, which indicates the minimum duration of viremia in this group, and there were generally no cases of deterioration in well-being with the development of critical conditions requiring oxygenation.
  A statistically significant difference was found between the indicators at admission and after 4-5 days between the control and experimental groups in terms of quantitative indicators of C reactive protein.

CONTACTS AND LOCATIONS:
Overall Officials: Erkin Musabaev, Professor, Study Chair — Rersearch Institute of Virology
Locations (1):
- Erkin Musabaev, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tempestilli M, Caputi P, Avataneo V, Notari S, Forini O, Scorzolini L, Marchioni L, Ascoli Bartoli T, Castilletti C, Lalle E, Capobianchi MR, Nicastri E, D'Avolio A, Ippolito G, Agrati C; COVID 19 INMI Study Group. Pharmacokinetics of remdesivir and GS-441524 in two critically ill patients who recovered from COVID-19. J Antimicrob Chemother. 2020 Oct 1;75(10):2977-2980. doi: 10.1093/jac/dkaa239. PMID 32607555
- [Background] Zu ZY, Jiang MD, Xu PP, Chen W, Ni QQ, Lu GM, Zhang LJ. Coronavirus Disease 2019 (COVID-19): A Perspective from China. Radiology. 2020 Aug;296(2):E15-E25. doi: 10.1148/radiol.2020200490. Epub 2020 Feb 21. PMID 32083985